CLINICAL TRIAL: NCT06401070
Title: Effect of Auricular Press Needle on Improvement of Patient Health Questionnaire-9 (PHQ-9) and Heart Rate Variability (HRV) Patient With Depression Symptoms in Chronic Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Nur Khasanah, Indonesia University, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DP.04.03
Record Dates: First submitted 2024-05-02; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Depression Symptoms; Chronic Pain
Keywords: acupuncture; auricular acupuncture; ear acupuncture; depression symptoms; chronic pain; press needle
MeSH Terms: conditions — Depression; Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): The control group was given a placebo press needle acupuncture (using plaster)
  Interventions: Device: Plesterin
- Intervention Group (Experimental): The intervention group was given press needle acupuncture
  Interventions: Device: Press needle acupuncture

INTERVENTIONS:
Device: Plesterin — The plaster used is a round plaster that resembles the shape of an acupuncture press needle.
  Arms: Control group
Device: Press needle acupuncture — Press needle acupuncture is a modality of acupuncture using tiny and very thin needles.
  Arms: Intervention Group

SUMMARY:
Depression is characterized by behavioral, cognitive and emotional changes. Depression can have a negative impact on decreasing quality of life because in many cases it occurs long-term. Chronic pain is often accompanied by various mental disorders, of which depression is the most common accompanying mental disorder. Chronic pain and depression themselves influence each other and are closely related, with globally around 30% to 45% of patients with chronic pain present with depression, and around 52% to 65% patients with depression suffer from chronic pain.

There are various therapeutic options for treating depression that aim to shorten depressive episodes and relieve symptoms. Multimodal therapy is needed in treating depression with chronic pain because there are biopsychosocial aspects involved. Pharmacological therapy has long-term side effects and the risk of drug dependence. Apart from that, depression patients with chronic pain, often receive pharmacological therapy such as non-steroidal anti-inflammatory drugs (NSAIDs) and opioids where the side effects and risk of drug dependence are higher. Therefore, it is necessary to choose a therapeutic modality that is relatively safe and effective in treating depression in chronic pain. In various studies it has been proven that acupuncture is an efficient and safe therapy for chronic pain patients with depression. Auricular acupuncture using pr ess needles has minimal pain and can be applied longer on acupuncture points.

This study aimed to assess the effectiveness of the auricular needle press on Patient with Depression Symptoms in Chronic Pain. This study was a double-blinded randomized clinical trial and was carried out on outpatients at Dr. Cipto Mangunkusumo National General Hospital Jakarta and Soerojo Hospital Magelang. There's also a collaborative study between the medical acupuncture department and the psychiatry department.

This study includes 60 participants who will be randomly allocated into 2 groups, the press needle and sham press needle groups. The press needles will be placed at 6 auricular points bilaterally : MA-TF1 Shenmen, MA-IC7 Heart, and MA-IT1 Cingulate gyrus.

The outcomes that will be assessed in this study are Patient Health Questionnaire-9 (PHQ-9) score and Heart Rate Variability (HRV).

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18-59 years.
* Subjects who experience depression symptoms with chronic pain
* Subjects with VAS >= 30 mm and < 70 mm from 100 mm during activity (daily activities or light exercise).
* Duration of pain > 3 months.
* Patient Health Questionnaire-9 Items (PHQ-9) score 5-19 on a scale of 0-27.
* Willing to take part in this study until completion and sign the informed consent.

Exclusion Criteria:

* Pain caused by malignancy.
* Patients diagnosed with major depression, depressive symptoms accompanied by psychotic symptoms, and depressive symptoms with antidepressant therapy.
* patients with medical emergencies or pregnancy.
* Infection, scar tissue, or malignancy at the acupuncture area.
* Anatomical abnormalities in the ear shape.
* Having hypersensitivity reaction to previous acupuncture therapy (metal allergy, atopy, keloid, or other skin hypersensitivity).
* Patients with cognitive impairment or impaired consciousness.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | before intervention, the first day, seventh day, and fourteenth-day post intervention
  Consists of nine questions that correspond to the nine questions of the diagnostic criteria for major depressive disorder of the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V). In each area assessed, there is a rating from 0 to 3 based on increasing frequency of difficulties. PHQ-9 scoring uses a 4-point Likert scale: 0 = "Not at all," 1 = "Some days," 2 = "More than half the days," and 3 = "Almost every day." With a total score ranging from 0 to 27
Heart Rate Variability (HRV). | before intervention, the first day, seventh day, and fourteenth-day post intervention
  To measure cardiac autonomic dysfunction non-invasively. HRV can be interpreted as the variability of heart rate. Methods for measuring HRV are categorized as time domain, frequency domain, geometric, and nonlinear.

CONTACTS AND LOCATIONS:
Overall Officials: Nur Khasanah, Principal Investigator — Medical Faculty Universitas Indonesia